CLINICAL TRIAL: NCT06130384
Title: Pain Reduction With Topical Bromfenac Versus Artificial Tear After Intravitreal Injection.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, Sunir Garg MD, Retina Physician and Surgeon, Co-Director of Retina Research, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012475
Record Dates: First submitted 2021-02-10; First posted 2023-11-14 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Pain; Intravitreal Injection; Pain, Acute
MeSH Terms: conditions — Pain; Acute Pain

STUDY DESIGN:
Intervention Model Description: All patients will receive both bromfenac 0.09% in the study eye and artificial tears in the control eye. Patients will be randomized to determine whether their right or left eye is the study eye.
Who Masked: Participant, Care Provider
Masking Description: Patients will be masked. The assistant instilling the eyedrop will be masked to which eyedrop is used for each eye.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bromfenac 0.09% (Experimental): At the time of the injection, the first eye will be randomized to a drop of artificial tear or bromfenac 0.09% and the second eye will receive the other agent.
  Interventions: Drug: Use of bromfenac 0.09% to reduce intravitreal injection pain
- Artificial Tear (Placebo Comparator): At the time of the injection, the first eye will be randomized to a drop of artificial tear or bromfenac 0.09% and the second eye will receive the other agent.
  Interventions: Drug: Use of artificial tears to reduce intravitreal injection pain

INTERVENTIONS:
Drug: Use of bromfenac 0.09% to reduce intravitreal injection pain — The eyedrop (bromfenac) will be given to the assigned eye.
  Arms: Bromfenac 0.09%
Drug: Use of artificial tears to reduce intravitreal injection pain — The eyedrop (artificial tears) will be given to the assigned eye.
  Arms: Artificial Tear

SUMMARY:
The purpose of this prospective interventional study is to compare post-intravitreal injection pain between eyes receiving topical bromfenac versus artificial tears as an analgesic after intravitreal injection.

DETAILED DESCRIPTION:
This proposed study is a double-masked randomized trial of adult patients receiving bilateral intravitreal injections. Patient data from March 2021 to June 2022 will be collected. Patient pain perception, quantified using the Wong-Baker FACES and the short-form McGill Pain Questionnaire, will be utilized to compare post-intravitreal injection pain between eyes receiving pre-injection bromfenac 0.09% ophthalmic solution versus artificial tears.

ELIGIBILITY:
Inclusion criteria are:

* Current patient of the Wills Eye Hospital Retina Service including all Mid Atlantic Retina offices
* Clinical indication of bilateral intravitreal anti-vascular endothelial growth factor (VEGF) injection as determined by the treating retina specialist for diseases such as age-related macular degeneration, choroidal neovascularization, diabetic macular edema, diabetic retinopathy, macular edema. proliferative retinopathy, or macular edema associated with retina vein occlusion.
* Age greater than 18
* Patient's that have had at least three prior injections in each eye

Exclusion criteria are:

* Prior ocular surgery (non-cataract)
* Herpetic eye disease
* Uncontrolled uveitis
* Active conjunctivitis, keratitis or keratopathy
* Current unilateral use of prescription eye drops.
* Allergy to NSAID

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Change in post-injection pain at 5 minutes using the Short Form McGill Pain Questionnaire Present Pain Intensity score | Patients will be asked in the office for their pain rating 5 minutes after injection
  Patients will be asked to report their pain on the Short Form McGill Questionnaire Present Pain Intensity score, ranging from 0 to 5, in which 5 is the worst pain level.
Change in post-injection pain at 5 minutes using the Wong-Baker Faces pain scale | Patients will be asked in the office for their pain rating 5 minutes after injection
  Patients will be asked to report their pain on the Wong-Baker Faces pain scale, ranging from 0 through 10, in which 10 is the worst pain level.
Change in post-injection pain at 6 hours using the Short Form McGill Pain Questionnaire Present Pain Intensity score. | Patients will be called for their rating 6 hours after injection
  Patients will be asked to report their pain on the Short Form McGill Questionnaire Present Pain Intensity score, ranging from 0 to 5, in which 5 is the worst pain level.
Change in post-injection pain at 5 minutes using the Wong-Baker Faces pain scale | Patients will be called for their rating 6 hours after injection
  from 0 through 10, in which 10 is the worst pain level.
Change in post-injection pain at 24 hours using the Short Form McGill Pain Questionnaire Present Pain Intensity score. | Patients will be called for their rating 24 hours after injection
  Patients will be asked to report their pain on the Short Form McGill Pain Questionnaire Present Pain Intensity score, ranging from 0 to 5, in which 5 is the worst pain level.
Change in post-injection pain at 5 minutes using the Wong-Baker Faces pain scale | Patients will be called for their rating 24 hours after injection
  from 0 through 10, in which 10 is the worst pain level.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Mid Atlantic Retina, Bethlehem, Pennsylvania
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Retina Consultants of San Antonio, San Antonio, Texas
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified data will be shared amongst researchers.
Supporting Information: Study Protocol, ICF